CLINICAL TRIAL: NCT06962345
Title: Changes in the Impact of Genitourinary Syndrome of Menopause With a Novel Nonhormonal Vulvovaginal Gel Assessed by PROMs. Phase 2, Single Arm, Interventional, Longitudinal, Clinical Trial. Part of STOP GSM PROJECT.
Brief Title: Changes in the Impact of Genitourinary Syndrome of Menopause With a Novel Nonhormonal Vulvovaginal Gel Assessed by PROMs.
Acronym: STOPGSMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mucosa Innovations, S.L. (Industry)
Collaborators: Hospital de La Luz (Other); Hospital Universitario Fundación Jiménez Díaz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STOPGSM01
Record Dates: First submitted 2025-04-29; First posted 2025-05-08 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Vulvar Atrophy; Vulvovaginal Signs and Symptoms; Genitourinary Syndrome of Menopause; Quality of Life; Menopause Related Conditions; Dyspareunia; Urinary Incontinence, Urgency-frequency; Sexual Function; Women´s Health; Vaginal Dryness
Keywords: Genitourinary Syndrome of Menopause; Vulvovaginal Signs and Symptoms; Patient Reported Outcome Measures; Quality of Life; Day-to-Day Impact of Vaginal Ageing; Women´s Health
MeSH Terms: conditions — Dyspareunia; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients diagnosed with Genitourinary Syndrome of Menopause. (Experimental): Patients diagnosed with Genitourinary Syndrome of Menopause using a non-hormonal vulvovaginal gel with tested composition XCMIM20m and PROMs questionnaire.
  Interventions: Device: Hormone-free vulvovaginal gel with the tested composition XCMIM20m

INTERVENTIONS:
Device: Hormone-free vulvovaginal gel with the tested composition XCMIM20m — Management of GSM in post-menopausal women will be measured with the combination of the application of the hormone-free vulvovaginal gel along the 8 weeks of the study and the use of a PROMs questionnaire. PROMS questionnaire will be delivered to the women at baseline and at the end of the study. Daily living quality of life domains of "activities of daily living", "emotional well-being", "sexual functioning", "self-perception and body image" will be evaluated.

SUMMARY:
The goal of this clinical trial is to improve the management of Genitourinary syndrome of menopause (GSM) to preliminary assess safety and effectivity of a novel hormone-free mucosa composition (XCMIM20m) applied topically to the vulvovaginal area. Symptoms of vaginal atrophy will be compared before and after 8 weeks of use of the tested gel with the Day-to-Day Impact of Vaginal Aging (DIVA) PROMs questionnaire to assess changes impact of GSM symptoms.

DETAILED DESCRIPTION:
The high prevalence of the Genitourinary Syndrome of the Menopause (GSM) previously known as vulvovaginal atrophy, atrophic vaginitis or urogenital atrophy, does not correlate with the fact that up until today GSM is still hugely underreported, underdiscussed, underdiagnosed as well as undertreated.

Postmenopausal women suffering from symptoms of GSM will be recruited after a routine visit at a Women's Unit at a General Hospital. The participants will self-assess their symptoms with the use of the Day-to-Day impact of Vaginal Aging (DIVA) questionnaire at baseline and after 8 weeks of use of the tested product. Self-assessment with PROMs will allow to obtain a greater knowledge of the physical and emotional state of patients as well as to deliver valuable information to women.

Criteria for a successful outcome will be if the use of the hormone-free agent is well accepted and if symptoms and quality of life improve after 8 weeks of intervention.

Daily dosage of XCMIM20m ((2-(trimethylazaniumyl) acetate; (2R,3R,4S)-pentane-1,2,3,4,5-pentol; Hexadecanoic acid; (9Z, 12Z)-octadeca-9,12-dienoic acid; octadecanoic acid; (Z)-hexadec-9-enoic acid; (Z)-octadec-9-enoic acid)) will be 2 ml of total product, divided in two applications of 1 ml every 12 hours, preferably morning and bedtime. To be spread topically onto the vulvar area, including the vaginal introitus. The gel will be further applied before sexual intercourse. No intravaginal applicator will be used as the agent will be manually applied directly onto the vulvar area from a 50 ml airless pump dispenser. Four pump applications from the pump dispenser are equivalent to 1ml of tested gel.

Adverse effects, such as allergic reaction, skin irritation, itching, discomfort, yeast infection, or any other, will be collected and if so, a detailed description and follow-up of the problem will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Patient has to have at least one symptom of GSM or suffer from symptoms related to vulvovaginal atrophy (as evidenced by gynecological examination with a Vaginal Health Index ≤15).
* Patient must be postmenopausal with at least 1 year without a menstrual period.
* Patient must consider that her quality of life is affected by GSM symptoms
* Patient not followed due to any gynecological disease.
* All participants must be able to understand and to fill in the self-reported questionnaires.

Exclusion Criteria:

* Patients that do not want to fill the questionnaire, especially the questions that address sexual functioning.
* Participants that use any oral products containing hormones or estrogen receptor modulators for the past 8 weeks, nor vaginal topical hormone products within 4 weeks, neither prescription nor non-prescription therapies for GSM, including topical vaginal non-hormonal lubricants or moisturizers for the last week.
* Patients with history of vulvar, vaginal and/or cervical malignancy.
* Patients having received radiotherapy treatment in the pelvic and/or genital region.
* Patients with any type of disease that causes alteration of collagenogenesis.
* Patients that use cytotoxic drugs leading to mucositis and alterations of tissue regeneration in the last 6 months.
* Patients having received laser and/or radiofrequency treatment for handling genital atrophy or other pelvic floor dysfunctions.
* Patients with active urinary and/or genital tract infection.
* Patients with history of malignant neoplasm of the urinary system.
* Patients with severe stress urinary incontinence (Sandvik test score equal to or greater than 8).
* Patients with diagnosis of pelvic organ prolapse grade III or higher according to the POP-Q classification.
* Patients with medical or surgery history that, at the investigator's discretion, does not allow participation in the study.
* Patients with any other condition that, at the investigator's discretion, implies that the patient is unable to understand the implication of participating in the study and/or following the established procedures.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Changes in GSM symptoms impact on quality of life domains after the intervention | Eight weeks of use of the tested product.
  Difference of magnitude of complaint by domain after 8 weeks of use of the tested product compared with baseline with the use of the PROMs questionnaire.
  The PROMs questionnaire will be the 23-item DIVA questionnaire comprising four domain scales: activities of daily living; emotional well-being; sexual functioning; and self-concept and body image.
  Each 23 items will be scored from 0 (meaning lowest impact/best quality of life) to 4 (meaning highest impact/worst quality of life).
  Total scores domain by domain will be assessed by calculating the average of scores for each item; higher scores will be interpreted as greater impact of GSM symptoms on women's quality of life and adscribed to each domain.

SECONDARY OUTCOMES:
Changes in the most affected women's quality of life domain after the intervention | Eight weeks of use of the tested product.
  Comparison in number of answers obtained for each score (0 to 4), domain by domain, at baseline and after 8 weeks of the use of the tested product assessed by the PROMs questionnaire.
  The PROMs questionnaire will be the 23-item DIVA questionnaire comprising four domain scales: activities of daily living; emotional well-being; sexual functioning; and self-concept and body image.
  Each 23 items will be scored from 0 (meaning lowest impact/best quality of life) to 4 (meaning highest impact/worst quality of life).
  Total scores domain by domain will be assessed by calculating the average of scores for each item; higher scores will be interpreted as greater impact of GSM symptoms on women's quality of life and adscribed to each domain.

OTHER OUTCOMES:
Adherence/compliance to the treatment | Eight weeks of use of the tested product.
  Adherence/compliance will be rated as good or poor.
  Adherence/compliance will be considered Good when the participant finishes the study period and fills in the second DIVA Questionnaire, and asks for extra product refill during the intervention and/or at the end of the intervention period.
  Adherence/compliance will be considered Poor when the participant does not finish the study period and/or does not fill in the second DIVA Questionnaire, and/or does not ask for any extra product refill during the intervention and/or at the end of the intervention period.
Changes in 23 items related to GSM symptoms impact on quality of life after the intervention | Eight weeks of use of the tested product
  Difference of intensity of each 23 complaints after 8 weeks of use of the tested product compared with baseline as described in the PROMs questionnaire. The PROMs questionnaire will be the 23-item DIVA questionnaire comprising four domain scales: activities of daily living; emotional well-being; sexual functioning; and self-concept and body image.
  Each 23 items will be scored from 0 (meaning lowest impact/best quality of life) to 4 (meaning highest impact/worst quality of life). Higher complaint scores will be interpreted as greater impact of GSM symptoms on women's quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Albi, MD, PhD, Principal Investigator — Hospital La Luz
Locations (1):
- Mucosa Innovations S.L., Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Portman DJ, Gass ML; Vulvovaginal Atrophy Terminology Consensus Conference Panel. Genitourinary syndrome of menopause: new terminology for vulvovaginal atrophy from the International Society for the Study of Women's Sexual Health and the North American Menopause Society. Menopause. 2014 Oct;21(10):1063-8. doi: 10.1097/GME.0000000000000329. PMID 25160739
- [Background] Management of symptomatic vulvovaginal atrophy: 2013 position statement of The North American Menopause Society. Menopause. 2013 Sep;20(9):888-902; quiz 903-4. doi: 10.1097/GME.0b013e3182a122c2. PMID 23985562
- [Background] Huang AJ, Gregorich SE, Kuppermann M, Nakagawa S, Van Den Eeden SK, Brown JS, Richter HE, Walter LC, Thom D, Stewart AL. Day-to-Day Impact of Vaginal Aging questionnaire: a multidimensional measure of the impact of vaginal symptoms on functioning and well-being in postmenopausal women. Menopause. 2015 Feb;22(2):144-54. doi: 10.1097/GME.0000000000000281. PMID 24983271
- [Background] Moral E, Delgado JL, Carmona F, Caballero B, Guillan C, Gonzalez PM, Suarez-Almarza J, Velasco-Ortega S, Nieto C; as the writing group of the GENISSE study. Genitourinary syndrome of menopause. Prevalence and quality of life in Spanish postmenopausal women. The GENISSE study. Climacteric. 2018 Apr;21(2):167-173. doi: 10.1080/13697137.2017.1421921. Epub 2018 Feb 7. PMID 29411644